CLINICAL TRIAL: NCT05873179
Title: Effects on Emphathy in Physiotherapy Students After Simulation With Kirkpatric Evaluation as an Active Method for Learning the Clinical Enterview
Brief Title: Effects on Emphathy in Physiotherapy Students After Simulation as an Active Method for Learning the Clinical Enterview
Status: Completed | Type: Observational
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, profesor, Universidad Complutense de Madrid
Other Study IDs: 23/29302
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Students
Keywords: Medical education; nursing education; physiotherapy; empathy
MeSH Terms: interventions — Role Playing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Role-playing for learning the clinical interview
  Interventions: Other: role-playing for learning the clinical interview

INTERVENTIONS:
Other: role-playing for learning the clinical interview — role-playing for learning the clinical interview

SUMMARY:
The aim of the main study is to find out the effects on empathy in physiotherapy students after role playing in the learning of the clinical history.

DETAILED DESCRIPTION:
Thirty-one first-year physiotherapy students will carry out the role-playing methodology to learn how to take a clinical history in physiotherapy.

Before and after the realization, they will be measured by means of a validated questionnaire in Spanish, the language in which they study, the variable of empathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are studying the first year of Physiotherapy at the Complutense University of Madrid and wish to participate in the study.

Exclusion Criteria:

* Students who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women who are studying the first year of Physiotherapy at the Complutense University of Madrid and wish to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-09-16 (Actual)

PRIMARY OUTCOMES:
Jefferson Scale or Medical Empathy Scale before role playing | Through study completion, an average of 1 week
  To determine the empathy levels of nursing students, the validated Jefferson Empathy Scale for health professions students will be used. This scale consists of 20 items, each of which is assessed using a seven-point Likert-type response scale (from 1 = 'strongly disagree' to 7 = 'strongly agree'). These items are divided into three subscales: 'perspective taking' (11 items), which refers to the cognitive aspects of empathy; 'compassionate care' (6 items), which is characterised by a combination of cognitive and affective aspects of empathy; and 'putting oneself in the patient's shoes' (three items), considered the inverse of emotional distancing . Ten of these items are positively worded, while the other 10 are negatively worded and should be reversed. The total scores range from 20 to 140 points. Higher scores reflect higher levels of empathy.
Empathy Quotent before role playing. | Through study completion, an average of 1 week
  It consists of 60 items, 40 measuring empathy and 20 control measures. Scores range from 0 to 80. It measures cognitive and affective empathy in adults. Equalizer allows classification into four categories, which facilitates comparison between groups. The cut-off for each level is: from 0 to 32 scores: low empathy (average scores in Asperger Syndrome is 20), from 33 to 52 scores: average empathy (average in men 42, average in women 47), from 53 to 63 scores: above average, from 64 to 80 scores: high empathy
Jefferson Scale or Medical Empathy Scale after role playing | Through study completion, an average of 1 week
  To determine the empathy levels of nursing students, the validated Jefferson Empathy Scale for health professions students will be used. This scale consists of 20 items, each of which is assessed using a seven-point Likert-type response scale (from 1 = 'strongly disagree' to 7 = 'strongly agree'). These items are divided into three subscales: 'perspective taking' (11 items), which refers to the cognitive aspects of empathy; 'compassionate care' (6 items), which is characterised by a combination of cognitive and affective aspects of empathy; and 'putting oneself in the patient's shoes' (three items), considered the inverse of emotional distancing . Ten of these items are positively worded, while the other 10 are negatively worded and should be reversed. The total scores range from 20 to 140 points. Higher scores reflect higher levels of empathy.
Empathy Quotent after role playing | Through study completion, an average of 1 week
  This questionnaire has been widely used to measure empathy in health science students.13 It consists of 60 items, 40 measuring empathy and 20 control measures. Scores range from 0 to 80. It measures cognitive and affective empathy in adults. Equalizer allows classification into four categories, which facilitates comparison between groups. The cut-off for each level is: from 0 to 32 scores: low empathy (average scores in Asperger Syndrome is 20), from 33 to 52 scores: average empathy (average in men 42, average in women 47), from 53 to 63 scores: above average, from 64 to 80 scores: high empathy.

CONTACTS AND LOCATIONS:
Locations (1):
- Eva María Martínez-Jimenez, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No